CLINICAL TRIAL: NCT04897737
Title: Study of the Feasibility and Acceptability of an Adherence Promotion Package for Postpartum Women on Pre-exposure Prophylaxis (PrEP)
Brief Title: Postpartum Pre-exposure Prophylaxis (PrEP) Study to Evaluate an Adherence Promotion Package for Postpartum Women on PrEP
Acronym: PPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K01TW011187-2; K01TW011187 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: HIV-1-infection
Keywords: PrEP; PMTCT; adherence; pregnant; postpartum; counseling; HIV self-testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): HIV self-testing kits and counseling on use for participant and partner use + enhanced adherence counseling including urine tenofovir test to provide biofeedback in women using PrEP
  Interventions: Behavioral: HIVST and enhanced adherence biofeedback; Diagnostic Test: Orasure/UrSure test
- Control (No Intervention): Standard of care intervention including facility based HIV testing, referral for partner to attend facility for testing, and PrEP adherence counseling without biofeedback

INTERVENTIONS:
Behavioral: HIVST and enhanced adherence biofeedback — The intervention includes the provision of an OraQuick HIV self-test (HIVST) for the woman and one test for each of her reported sex partners, along with instructions on how to use and interpret the results. Women were asked to report back within one month if their partner was able to test via a SMS, WhatsApp or by bringing in the test to confirm that he had tested.
  Women then received adherence based feedback following the urine lateral flow assay (that measures recent tenofovir use in past 48 hours). Study counsellors requested that women provide a urine sample that was tested using the UrSure/Orasure test that provides feedback on the result in 2-3 minutes. Counselors provided counseling based on the results including how to improve daily adherence (for women without tenofovir present in their urine) and importance of condom use.
  Other Names: urine tenofovir test; HIV self test
  Arms: Intervention
Diagnostic Test: Orasure/UrSure test — See above
  Other Names: urine tenofovir test
  Arms: Intervention

SUMMARY:
The postpartum PrEP study (PPS) seeks to evaluate how best to improve adherence to PrEP in postpartum women and to evaluate how acceptable it is to offer HIV self tests for the participant and partner, and provide enhanced adherence biofeedback following a urine test of recent PrEP use (measuring tenofovir). The primary outcome is recent PrEP adherence following the intervention. The secondary outcome is HIV testing uptake in participants' partners.

DETAILED DESCRIPTION:
Pregnant and breastfeeding women in South Africa are at very high risk of HIV acquisition and vertical HIV transmission during pregnancy, labour and breastfeeding. One-third to half of perinatal HIV transmission occurs in women who are seroconvert during the pregnancy and post-partum period. Effective use of pre-exposure prophylaxis (PrEP) could contribute to eliminating maternal HIV acquisition, and hence mother to child transmission (MTCT) of HIV. However, PrEP efficacy requires high levels of adherence, and adherence requires high levels of acceptability, yet there are few data on how best to promote adherence to PrEP in postpartum women.

We will conduct a study of the feasibility and acceptability of an adherence promotion package in n=100 postpartum women enrolled in an ongoing PrEP study (PrEP-PP; ongoing, R01MH116771) to evaluate the feasibility, acceptability and efficacy of a package of interventions to improve PrEP adherence in pregnancy and postpartum women. Specifically the package of interventions will include:

* Offer of HIV self-test in women and their partners with counseling on use
* Integrating urine based lateral flow assays in enhanced counseling using biofeedback on adherence levels to postpartum women on PrEP

The primary outcome is recent PrEP adherence at 1-month following the intervention. The secondary outcome is HIV testing uptake in participants' partners.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in PrEP-PP study and on PrEP
2. 18+ years old
3. confirmed HIV-negative (confirmed with a 4th generation antigen HIV test)
4. confirmed to be postpartum (1-6 months postpartum)
5. confirmed to currently have a male partner
6. confirmed to have a cell phone that can read and respond to SMS/Whatsapp messages

Exclusion Criteria:

Failure to meet all of inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gugulethu Midwife Obstetric Unit, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Researchers can contact PI to decide on sharing IPD for further analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: To contact PI for access to study data

REFERENCES:
- [Result] Joseph Davey DL, Dovel K, Mvududu R, Nyemba D, Mashele N, Bekker LG, Gorbach PM, Coates TJ, Myer L. Pre-exposure Prophylaxis Recent Adherence With Real-Time Adherence Feedback and Partner Human Immunodeficiency Virus Self-Testing: A Pilot Trial Among Postpartum Women. Open Forum Infect Dis. 2021 Dec 23;9(2):ofab609. doi: 10.1093/ofid/ofab609. eCollection 2022 Feb. PMID 35097151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2020 and April 2021, trained study staff recruited cisgender women from the PrEP-PP cohort for the pilot study. Eligibility criteria included having given birth to a live infant in the preceding 4-24 weeks, documented HIV-negative status in the study on the date of screening, initiating PrEP in the recently completed pregnancy, and reported having at least 1 sexual partner.
Groups:
- Intervention: HIV self-testing kits and counseling on use for participant and partner use + enhanced adherence counseling including urine tenofovir test to provide biofeedback in women using PrEP
  HIVST and enhanced adherence biofeedback: The intervention includes the provision of an OraQuick HIV self-test (HIVST) for the woman and one test for each of her reported sex partners, along with instructions on how to use and interpret the results. Women were asked to report back within one month if their partner was able to test via a SMS, WhatsApp or by bringing in the test to confirm that he had tested.
  Women then received adherence based feedback following the urine lateral flow assay (that measures recent tenofovir use in past 48 hours). Study counsellors requested that women provide a urine sample that was tested using the UrSure/Orasure test that provides feedback on the result in 2-3 minutes. Counselors provided counseling based on the results including how to improve daily adherence (for women without tenofovir present in their urine) and importance of condom use.
  Orasure/UrSure test: See above
Period: Overall Study
Arm/Group | Intervention | Control
Started | 53 | 53
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 53 | 106
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 26 [23 to 31] | 26 [23 to 31] | 26 [23 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 53 | 106
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Recent PrEP Adherence
Description: The primary study outcome is recent PrEP adherence according to urine tenofovir test by study arm.
Time Frame: 1 month after intervention
Population: Postpartum women on PrEP who had urine tenofovir present in urine (indicative of taking PrEP in last 2-3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 53
Participants | 33 | 18
Statistical Analysis 1: Comparison: Intervention vs Control; All analyses were by intention-to-treat. In the case of missing outcomes for participants who did not return for the follow-up visit, we assigned outcome values of the following: poor PrEP adherence (TFV undetected) and partner not tested for HIV. We constructed univariate Poisson regression models with robust standard errors to examine the predictors of outcomes of interests. Model results are presented as crude risk ratios (RRs) and risk differences (RDs) with 95% CIs; Test type: Superiority; p < 0.001, Mixed Models Analysis; Risk Ratio (RR) = 1.83, 95% CI 2-sided [1.19 to 2.82]

2. Secondary Outcome: Participant Partners Who Tested for HIV
Description: The secondary outcome was number of partners who tested for HIV (as reported by the female partner and confirmed with photo or used HIVST in intervention arm) by study arm.
Time Frame: 1 month after intervention
Population: Postpartum women on PrEP
Measure: Number; unit: male partners
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 53
male partners | 35 | 9
Statistical Analysis 1: Comparison: Intervention vs Control; All analyses were by intention-to-treat. In the case of missing outcomes for participants who did not return for the follow-up visit, we assigned outcome values of the following: poor PrEP adherence (TFV undetected) and partner not tested for HIV. We constructed univariate Poisson regression models with robust standard errors to examine the predictors of outcomes of interests. Model results are presented as crude risk ratios (RRs) and 95% CIs; Test type: Superiority; p < 0.001, Regression, Linear; Risk Ratio (RR) = 3.89, 95% CI 2-sided [2.08 to 7.27]; RD=49.1% (95% CI=32.8, 65.3), p<0.001

3. Other Pre Specified Outcome: Adverse Events
Description: Any adverse event occurring in the study including intimate partner violence, relationship issues, or conflict
Time Frame: During study monitoring
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Any adverse event including intimate partner violence (IPV) as defined by WHO
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 1/53 | 0/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=53) | Control (N=53)
Intimate Partner Violence (Psychiatric disorders) | 1 (1) | 0 (0) — Partner yelling and conflict after testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT04897737/Prot_SAP_000.pdf